CLINICAL TRIAL: NCT00055666
Title: Compassionate Use Of Oral Beclomethasone Dipropionate For Treatment Of Gastrointestinal Graft Versus Host Disease
Brief Title: Compassionate Use of Beclomethasone in Treating Patients With Graft-Versus-Host Disease of the Gastrointestinal Tract
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Philip McCarthy,, Roswell Park Cancer Institute
Allocation: Non-Randomized | Masking: None | Purpose: Supportive Care
Other Study IDs: CDR0000270747; RPCI-DS-01-04
Record Dates: First submitted 2003-03-06; First posted 2003-03-07 (Estimated); Last update posted 2011-03-08 (Estimated); Status verified 2011-03

CONDITIONS: Graft Versus Host Disease
Keywords: graft versus host disease
MeSH Terms: conditions — Graft vs Host Disease | interventions — Beclomethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: beclomethasone dipropionate

SUMMARY:
RATIONALE: Beclomethasone may be effective in treating patients who have graft-versus-host disease of the gastrointestinal tract.

PURPOSE: Compassionate use of beclomethasone in treating patients who have graft-versus-host disease of the gastrointestinal tract that has not responded to previous therapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Provide beclomethasone dipropionate to patients with gastrointestinal graft-versus-host disease refractory to standard therapy or with a contraindication to systemic steroids.
* Minimize the serious side effects associated with systemic steroid use in these patients.

OUTLINE: Patients receive oral beclomethasone dipropionate 4 times daily for 28 days in the absence of graft-versus-host disease progression or unacceptable toxicity. Patients may then receive a second course for 31 days if symptoms of graft-versus-host disease persist. Patients may receive up to 4 treatments (1 or 2 courses each) per year.

PROJECTED ACCRUAL: A total of 24-45 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Clinically or pathologically confirmed graft-versus-host disease of the gastrointestinal tract

  * Failed standard therapy with or has a contraindication to systemic immunosuppressive agents
* No clinically significant intestinal infection (confirmed by stool culture)
* No persistent vomiting of all oral intake
* Not a candidate for approved beclomethasone dipropionate Enteron Pharmaceuticals protocol

PATIENT CHARACTERISTICS:

Age

* 4 to 70

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* Able to swallow medication

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* See Disease Characteristics

Radiotherapy

* Not specified

Surgery

* Not specified

Ages: 4 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2001-03; Primary Completion 2005-02 (Actual); Study Completion 2006-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip L. McCarthy, MD, Study Chair — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States